CLINICAL TRIAL: NCT05044403
Title: Clinical Impact of Hemoperfusion With a Neutral Macroporous Resin Cartridge as Adjunctive Treatment in Septic Patients With Multiorgan Dysfunction Syndrome (MODS) Admitted to Intensive Care Units.
Brief Title: Hemoperfusion in Critical Patients With Septic Multiorgan Dysfunction Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hospital General Universitario de Castellón (Other); Hospital Universitario La Paz (Other); Hospital de Granollers (Other); Hospital General Universitario Santa Lucía (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUL-HEMO-2021-1
Record Dates: First submitted 2021-08-03; First posted 2021-09-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hemoperfusion; Multiorgan Failure; Sepsis
MeSH Terms: conditions — Multiple Organ Failure; Sepsis | interventions — Hemoperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment (Active Comparator): Patients receiving conventional treatment for multiorganic dysfunction syndrome from septic origin.
  Interventions: Procedure: Conventional treatment
- Extracorporeal support with haemoperfusion treatment (Experimental): Patients receiving extracorporeal support with haemoperfusion for multiorganic dysfunction syndrome from septic origin.
  Interventions: Procedure: Extracorporeal support with haemoperfusion

INTERVENTIONS:
Procedure: Extracorporeal support with haemoperfusion — Use of extracorporeal support with haemoperfusion
  Arms: Extracorporeal support with haemoperfusion treatment
Procedure: Conventional treatment — Conventional treatment
  Arms: Conventional treatment

SUMMARY:
Low-level interventional clinical trial to evaluate the effectiveness and safety of extracorporeal support with hemoperfusion in critical patients with septic multiorgan dysfunction syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a sepsis diagnosis, according to the diagnostic criteria of the International Sepsis-3 Consensus Conference, and without response to the treatment of septic shock who meet the following conditions:
* Sepsis of abdominal origin with controlled infectious focus.
* Noradrenaline dose> 0.5 µg / kg / min to maintain adequate organ perfusion after optimization of fluid therapy.
* Dysfunction of two or more organs with SOFA ≥ 9 (5).
* Blood lactate ≥ 2 mmol / L.
* Procalcitonin (PCT)> 10 ng / mL.
* CRP> 100 mg / L.
* IL-6> 2000 pg / ml.

Exclusion Criteria:

* Age under 18 years or over 80 years.
* Pregnancy or breastfeeding.
* Terminally ill patients or with a life expectancy of less than 48 hours.
* Thrombocytopenia <60,000 / mm3.
* Pancytopenia.
* Severe coagulopathy with high risk of bleeding.
* Inclusion in another research protocol.
* In case of re-entry during the study period, only the first admission will be included.
* Use of another haemoperfusion device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
IL-6 plasmatic concentration | During hemoperfusion
  Analyze the patient's variation of IL-6 plasmatic concentration during the hemoperfusion process
Adverse events | During hemoperfusion
  Analyze the presence of adverse events during the hemoperfusion process
Organ failure | During hemoperfusion
  Analyze the number and severity of failed organs during the hemoperfusion process
Vasopressors dose | During hemoperfusion
  Analyze the patient's vasopressor dose variation during the hemoperfusion process
Mean arterial pressure | During hemoperfusion
  Analyze the patient's variation of mean arterial pressure during hemoperfusion
Vasopressors dose | During ICU stay
  Analyze the number of days on vasopressor support during ICU stay
Mechanical ventilation | During ICU stay
  Analyze the number of days on mechanical ventilation during ICU stay
Renal replacement therapy | During ICU stay
  Analyze the number of days on renal replacement therapy during ICU stay
ICU length of stay | Post-Intensive Care Unit discharge
  Analyze the patient's length of stay in ICU
ICU survival | Post-Intensive Care Unit discharge
  Analyze the patient's survival in ICU
Hospital stay | post-hospital discharge
  Analyze the patient's length of stay post-Intensive Care Unit discharge
Hospital survival | Post-hospital discharge
  Analyze the patient's survival post-hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Sanchez Moran, Principal Investigator — Hospital General Universitario de Castellon
Locations (1):
- Hospital General Universitario de Castellon, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Background Abdominal sepsis remains a major challenge in critical care, often associated with high morbidity and mortality. Hemoadsorption therapy has been proposed as a strategy to modulate the systemic inflammatory response in septic patients. However, clinical evidence in the abdominal sepsis population is limited.
  Conclusions Haemoadsorption appears to be a feasible and safe intervention in patients with abdominal sepsis. Preliminary results suggest potential benefits in inflammatory modulation, organ function improvement, and mortality reduction. Larger, more robust clinical trials are required to confirm efficacy and clarify its impact on clinical outcomes. A more comprehensive and detailed analysis of the results will be provided upon completion of the study.